CLINICAL TRIAL: NCT06074835
Title: Automation of Gamete Preparation, Intracytoplasmic Sperm Injection (ICSI), Embryo Culture, and Vitrification: A Proof of Concept Study
Brief Title: Automation of Gamete Preparation, Intracytoplasmic Sperm Injection (ICSI), Embryo Culture, and Vitrification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Conceivable Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CP001
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Robot-assisted gamete preparation, ICSI, embryo culture and vitrification) (Experimental)
  Interventions: Device: Gamete preparation, ICSI, embryo culture and vitrification robot assistant
- Control group (routine manual ICSI workflow) (Active Comparator)
  Interventions: Other: Routine Manual ICSI Workflow

INTERVENTIONS:
Device: Gamete preparation, ICSI, embryo culture and vitrification robot assistant — Patients undergoing an assisted conception treatment with medical indication to perform ICSI may be recruited in this study. The study will follow a sibling-oocyte and/or sibling embryo study design where oocytes and/or embryos obtained from a specific patient or couple will be randomly distributed across two groups (test and control) and undergo one or more elements of an automated assisted conception laboratory workflow (for the test group) or a standard assisted conception laboratory workflow (for the control group). Before distributing the samples, an embryologist will slightly blur the vision of the samples so that their morphology can no longer be clearly assessed. Robotic automation may include any of the following steps: robotic sperm preparation, robotic oocyte selection and denudation, robotic sperm injection, automated embryo culture, and automated cryopreservation. The resulting embryos may be employed for embryo transfer.
  Arms: Test group (Robot-assisted gamete preparation, ICSI, embryo culture and vitrification)
Other: Routine Manual ICSI Workflow — Routine Manual Icsi Workflow
  Arms: Control group (routine manual ICSI workflow)

SUMMARY:
Patients suffering from infertility may seek assisted conception treatment. In a full treatment cycle, the sperm and eggs (gametes) from the intended parents will be looked after by skilled laboratory staff (embryologists) who will rely on manual laboratory processes to achieve fertilization. The most commonly employed method to achieve fertilization is intracytoplasmic sperm injection (ICSI), a treatment that involves the injection of a single sperm cell directly inside an egg. The embryos so obtained are then be maintained in an appropriate environment (incubator) for several days before deciding whether they can be immediately used to attempt to establish a pregnancy (embryo transfer), or should be frozen in preparation for a future treatment (cryopreservation).

The laboratory steps required to complete a full assisted conception treatment (from sperm and egg retrieval, to fertilization, and then to embryo transfer and/or cryopreservation) are often manual and time-consuming, and thus the success of the treatment is highly dependent on the skill of individual staff and outcomes can be affected by fatigue, stress, and workload.

The combination of robotics and artificial intelligence (AI) has the potential to provide improvements to, and standardize, the fertility laboratory, but such integration has not been achieved routinely. Other medical fields, such as regenerative medicine, have long benefited from the implementation of robotic solutions; however, modern automation has yet to find its way into the fertility laboratory.

The goal for Conceivable Life Sciences (the study sponsor) is the delivery of a suite of solutions that, collectively, will allow a fully autonomous ICSI cycle to take place (from sperm/egg preparation, to sperm injection, to embryo culture and cryopreservation) in an effort to reduce costs, assist laboratory staff, and possibly, improve outcomes. The purpose of this study is to deliver a core aspect of this project: the digital control and individual automation of all key steps of a complete laboratory workflow. The data generated in this study will help the future development of these automated systems.

Patients undergoing an ICSI treatment may be recruited in this study. Their gametes (sperm and/or eggs) may be distributed across two groups (test and control) and undergo one or more elements of an automated full assisted conception workflow (for the test group) or a standard assisted conception workflow (for the control group). Robotic automation may include any of the following steps: robotic sperm preparation, robotic oocyte selection and denudation, robotic sperm injection, automated embryo culture, and automated cryopreservation. The resulting embryos may be employed for embryo transfer.

The main hypothesis of this study is that the use of robotic assistants as part of a full assisted conception cycle may improve laboratory workflows without reducing the treatment success rates.

ELIGIBILITY:
Inclusion Criteria:

* Medical indication to perform ICSI.
* Informed consent signed by the patients before treatment.
* Medical indication for the use of autologous or donor oocytes.
* Medical indication for the use of autologous or donor sperm.
* Motile sperm.

Exclusion Criteria:

* Recurrent pregnancy loss.
* Previous history of total fertilization failure.
* Surgical sperm retrieval.
* Severe male factor infertility.
* Known semen liquefaction problems.
* Any other case abnormalities that could potentially reduce success rates according to the criteria of the senior embryologist in charge.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2025-10-04 (Actual)

PRIMARY OUTCOMES:
Timing | 6 weeks from enrolment
  Time to complete each automated procedure
Efficiency | 6 weeks from enrolment
  proportion of automated procedures achieving their goal
Autonomy | 6 weeks from enrolment
  proportion of completed procedure not requiring human intervention
Walk-away time | 6 weeks from enrolment
  time savings realized by an embryologist who is able to attend other duties while the robotic assistant is at work

SECONDARY OUTCOMES:
Sperm survival and quality (seminogram) | 6 weeks from enrolment
Proportion of oocytes fertilized | 6 weeks from enrolment
Embryos survival and quality (by morphology assessment) | 6 weeks from enrolment
Clinical pregnancy rates following embryo transfer | 8 weeks from enrolment
Live birth rates following embryo transfer | within 12 months of primary completion

CONTACTS AND LOCATIONS:
Locations (1):
- Hope Fertility Centre, Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures, and appendices).
  Data sharing is subject to ethical, legal, and privacy considerations. We are committed to following established guidelines and best practices for data sharing.
  This plan has been updated to provide more detailed information on access criteria.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal.
  Proposals may be submitted up to 36 months following article publication. Proposals should be directed to Jacques@Conceivable.life; to gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Chavez-Badiola A, Mendizabal-Ruiz G, Flores-Saiffe Farias A, Costa-Borges N, Murray A, Alikani M, Silvestri G, Millan C, Hernandez-Morales E, Valencia-Murillo R, Medina V, Mestres E, Valadez Aguilar A, Ocegueda-Hernandez V, Acosta-Gomez F, Alvarez Lopez A, Acacio M, Matia-Algue Q, Espinoza Figueroa JG, Campos Olmedo LM, Barragan CP, Sanchez-Gonzalez DJ, Cohen J. Automated oocyte retrieval, denudation, sperm preparation, and ICSI in the IVF laboratory: a proof-of-concept study and report of the first live births. Hum Reprod. 2025 Dec 26:deaf240. doi: 10.1093/humrep/deaf240. Online ahead of print. PMID 41453368